CLINICAL TRIAL: NCT05366023
Title: Elucidating the Necessary Components and Mechanisms of Cognitive Training
Brief Title: Elucidating the Necessary Active Components of Training
Acronym: ENACT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clemson University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Penn State University (Other); University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: U01AG062370 (NIH); U01AG062370 (NIH)
Record Dates: First submitted 2022-05-04; First posted 2022-05-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Alzheimer Disease; Cognitive Change; Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (20):
- No contact (No Intervention): 0 hours of activities during intervention period of study
- TDD1 (Experimental): 10 hours of top-down driven cognitive training games
  Interventions: Behavioral: TDD1
- TDD2 (Experimental): 10 hours of top-down driven cognitive training games
  Interventions: Behavioral: TDD2
- TDD1 + TDD2 (Experimental): 20 hours of top-down driven cognitive training games
  Interventions: Behavioral: TDD1; Behavioral: TDD2
- BUD1 (Experimental): 10 hours of bottom-up driven cognitive training games
  Interventions: Behavioral: BUD1
- BUD2 (Experimental): 10 hours of bottom-up driven cognitive training games
  Interventions: Behavioral: BUD2
- BUD1 + BUD2 (Experimental): 20 hours of bottom-up driven cognitive training games
  Interventions: Behavioral: BUD1; Behavioral: BUD2
- BUD2 + TDD2 (Experimental): 10 hours of bottom-up driven cognitive training games plus 10 hours of top-down driven cognitive training games
  Interventions: Behavioral: BUD2; Behavioral: TDD2
- BUD1 + TDD1 (Experimental): 10 hours of bottom-up driven cognitive training games plus 10 hours of top-down driven cognitive training games
  Interventions: Behavioral: BUD1; Behavioral: TDD1
- BUD2 + TDD1 (Experimental): 10 hours of bottom-up driven cognitive training games plus 10 hours of top-down driven cognitive training games
  Interventions: Behavioral: BUD2; Behavioral: TDD1
- BUD2 + TDD1 + TDD2 (Experimental): 10 hours of bottom-up driven cognitive training games plus 20 hours of top-down driven cognitive training games
  Interventions: Behavioral: BUD2; Behavioral: TDD1; Behavioral: TDD2
- BUD1 + TDD2 (Experimental): 10 hours of bottom-up driven cognitive training games plus 10 hours of top-down driven cognitive training games
  Interventions: Behavioral: BUD1; Behavioral: TDD2
- BUD1 + TDD1 + TDD2 (Experimental): 10 hours of bottom-up driven cognitive training games plus 20 hours of top-down driven cognitive training games
  Interventions: Behavioral: BUD1; Behavioral: TDD1; Behavioral: TDD2
- BUD1 + BUD2 + TDD2 (Experimental): 20 hours of bottom-up driven cognitive training games plus 10 hours of top-down driven cognitive training games
  Interventions: Behavioral: BUD1; Behavioral: BUD2; Behavioral: TDD2
- BUD1 + BUD2 + TDD1 (Experimental): 20 hours of bottom-up driven cognitive training games plus 10 hours of top-down driven cognitive training games
  Interventions: Behavioral: BUD1; Behavioral: BUD2; Behavioral: TDD1
- BUD1 + BUD2 + TDD1 + TDD2 (Experimental): 20 hours of bottom-up driven cognitive training games plus 20 hours of top-down driven cognitive training games
  Interventions: Behavioral: BUD1; Behavioral: BUD2; Behavioral: TDD1; Behavioral: TDD2
- CSA10 (Active Comparator): 10 hours of cognitive stimulating activities
  Interventions: Behavioral: CSA10
- CSA20 (Active Comparator): 20 hours of cognitive stimulating activities
  Interventions: Behavioral: CSA20
- CSA30 (Active Comparator): 30 hours of cognitive stimulating activities
  Interventions: Behavioral: CSA30
- CSA40 (Active Comparator): 40 hours of cognitive stimulating activities
  Interventions: Behavioral: CSA40

INTERVENTIONS:
Behavioral: BUD1 — 10 hours of bottom-up driven computerized cognitive training designed to improve processing speed and divided attention
  Arms: BUD1; BUD1 + BUD2; BUD1 + BUD2 + TDD1; BUD1 + BUD2 + TDD1 + TDD2; BUD1 + BUD2 + TDD2; BUD1 + TDD1; BUD1 + TDD1 + TDD2; BUD1 + TDD2
Behavioral: BUD2 — 10 hours of bottom-up driven computerized cognitive training designed to improve divided attention
  Arms: BUD1 + BUD2; BUD1 + BUD2 + TDD1; BUD1 + BUD2 + TDD1 + TDD2; BUD1 + BUD2 + TDD2; BUD2; BUD2 + TDD1; BUD2 + TDD1 + TDD2; BUD2 + TDD2
Behavioral: TDD1 — 10 hours of top-down driven computerized cognitive training designed to improve multiple object tracking
  Arms: BUD1 + BUD2 + TDD1; BUD1 + BUD2 + TDD1 + TDD2; BUD1 + TDD1; BUD1 + TDD1 + TDD2; BUD2 + TDD1; BUD2 + TDD1 + TDD2; TDD1; TDD1 + TDD2
Behavioral: TDD2 — 10 hours of top-down driven computerized cognitive training designed to improve executive function
  Arms: BUD1 + BUD2 + TDD1 + TDD2; BUD1 + BUD2 + TDD2; BUD1 + TDD1 + TDD2; BUD1 + TDD2; BUD2 + TDD1 + TDD2; BUD2 + TDD2; TDD1 + TDD2; TDD2
Behavioral: CSA10 — 10 hours of computerized games
  Arms: CSA10
Behavioral: CSA20 — 20 hours of computerized games
  Arms: CSA20
Behavioral: CSA30 — 30 hours of computerized games
  Arms: CSA30
Behavioral: CSA40 — 40 hours of computerized games
  Arms: CSA40

SUMMARY:
Loss of independence, cognitive decline, and difficulties in everyday function are areas of great concern for older adults and their families. Cognitive training is one low cost, noninvasive training intervention that has repeatedly demonstrated reliable transfer effects to maintained cognition, everyday function, health, and most recently, a 29% reduction in incident dementia. Importantly, many of these everyday function effects are maintained across five to ten years including: maintained driving mobility, 50% reduction in at-fault vehicle crashes, and maintained Instrumental Activities of Daily Living (IADL). Although clearly an important and effective intervention, the moderators and mechanisms underlying this program are unknown.

The overall objective in this planning grant is to lay the conceptual and methodological foundation to explore cognitive, psychosocial, lifestyle behaviors, and biomarker mechanisms and moderators of two forms of conceptually driven cognitive training. Additionally, this study will examine how cognitive and psychosocial factors within daily life account for the transfer of cognitive training to everyday function. We will use a factorial design to randomize adults ages 55-85 to 0, 10, 20, 30, or 40 hours of two forms of cognitive training, a combined training, or an active comparison condition (Phase 1). An additional sample of participants will complete 20 hours of two forms of cognitive training or the active comparison group as well as provide blood samples (Phase 2).

Across the study period, participants will complete cognitive, health, lifestyle, and psychosocial assessments at baseline, posttest, and approximately three month follow-up assessments in person or remotely using a study-provided laptop. Additionally, all participants will be asked to complete daily cognitive, health, lifestyle, and psychosocial measures daily using study-provided smartphones.

This study will allow us to test the feasibility of our enrollment, assessment and training protocols for a future multisite clinical trial. This exploratory study is the first of its kind and will be used to provide important data relevant to a future larger randomized controlled trial examining mediators of cognitive training in a representative sample of adults. This information will assist in the future development of more effective home- and community-based interventions that maintain everyday function.

ELIGIBILITY:
Inclusion Criteria:

* Phase 1:

  * Age 55-85 community-dwelling adults
  * Written informed consent obtained
  * No reported evidence of or diagnosis of dementia/Alzheimer's Disease; score of 5 or greater on the MIS-t administered during phone screening
  * Willing and able to participate in the up to 9 months of the study duration
  * Is proficient in written and spoken English
* Phase 2:

  * All Phase 1 criteria plus willingness and ability to provide two blood samples at baseline and posttest

Exclusion Criteria:

* Phase 1 exclusions:

  * Failure to meet any of the above eligibility criteria
  * Use of video games for more than 2 hours/week over the previous 2 years
  * Currently engaged in a cognitive program such as Brain HQ or Lumosity
* Phase 2 exclusion:

In addition to Phase 1 exclusion, also criteria below:

• Inability or unwillingness to travel to Clemson to provide two in-person blood samples at baseline and posttest

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2022-02-21 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Protocol compliance | Baseline through 3 month follow-up visit
  Participants complete laptop and phone activities as outlined in the study protocol

SECONDARY OUTCOMES:
Complex Instrumental Activities of Daily Living | Baseline through 3 month follow-up visit
  Measures of everyday functioning as detailed in the study protocol

CONTACTS AND LOCATIONS:
Locations (1):
- Clemson University Institute for Engaged Aging, Seneca, South Carolina, United States